CLINICAL TRIAL: NCT06057103
Title: A Study to Evaluate Drug-drug Interaction of ZX-7101A Tablets and Oseltamivir Phosphate Capsules in Healthy Adult Subjects -a Single-center, Open-labelled, Six-sequence, Three-cycle Crossover Design
Brief Title: A Study to Evaluate Drug-drug Interaction of ZX-7101A Tablets and Oseltamivir Phosphate Capsules in Healthy Adult Subjects
Acronym: ZX-7101A-208
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Nanjing Zenshine Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: ZX-7101A-208
Record Dates: First submitted 2023-09-12; First posted 2023-09-28 (Actual); Last update posted 2024-11-04 (Actual); Status verified 2024-10

CONDITIONS: Drug Interaction
MeSH Terms: interventions — Oseltamivir

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (6):
- ZX-7101A-1 (Other)
  Interventions: Drug: ZX-7101A; Drug: Oseltamivir; Drug: ZX-7101A and Oseltamivir
- ZX-7101A-2 (Other)
  Interventions: Drug: ZX-7101A; Drug: ZX-7101A and Oseltamivir; Drug: Oseltamivir
- Oseltamivir-1 (Other)
  Interventions: Drug: Oseltamivir; Drug: ZX-7101A; Drug: ZX-7101A and Oseltamivir
- Oseltamivir-2 (Other)
  Interventions: Drug: Oseltamivir; Drug: ZX-7101A and Oseltamivir; Drug: ZX-7101A
- Combined-1 (Other)
  Interventions: Drug: ZX-7101A and Oseltamivir; Drug: ZX-7101A; Drug: Oseltamivir
- Combined-2 (Other)
  Interventions: Drug: ZX-7101A and Oseltamivir; Drug: Oseltamivir; Drug: ZX-7101A

INTERVENTIONS:
Drug: ZX-7101A — ZX-7101A Tablets single dose tablet, 80 mg, Oral
  Arms: ZX-7101A-1; ZX-7101A-2
Drug: Oseltamivir — Oseltamivir phosphate capsule was administered as a single drug, 75 mg twice daily, for 5 days,Oral
  Arms: Oseltamivir-1; Oseltamivir-2; ZX-7101A-1
Drug: ZX-7101A and Oseltamivir — ZX-7101A tablet (80mg, single dose) was combined with oseltamivir phosphate capsule (75 mg twice daily),Oral
  Arms: Combined-1; Combined-2; Oseltamivir-2; ZX-7101A-1; ZX-7101A-2
Drug: ZX-7101A — ZX-7101A Tablets single dose tablet, 80 mg, Oral
  Arms: Combined-1; Oseltamivir-1; Oseltamivir-2
Drug: Oseltamivir — Oseltamivir phosphate capsule was administered as a single drug, 75 mg twice daily, for 5 days,Oral
  Arms: Combined-1; Combined-2; ZX-7101A-2
Drug: ZX-7101A and Oseltamivir — ZX-7101A tablet (80mg, single dose) was combined with oseltamivir phosphate capsule (75 mg twice daily),Oral
  Arms: Oseltamivir-1
Drug: ZX-7101A — ZX-7101A Tablets single dose tablet, 80 mg, Oral
  Arms: Combined-2

SUMMARY:
The primary object of this study is evaluating the effect of multiple oral oseltamivir phosphate capsules on the pharmacokinetic profile of the active metabolite ZX-7101 after a single oral administration of ZX-7101A tablet in healthy Chinese adult subjects.

The seongdary object is evaluating combined or uncombined multiple oral oseltamivir phosphate in healthy Chinese adult subjects.

ELIGIBILITY:
Inclusion Criteria:

Healthy male or female subjects between the ages of 18 and 45 years (including the threshold value, based on the date of signing ICF).

Weight: Male weight ≥50 kg, female weight ≥45 kg, BMI between 19.0 and 28.0 kg/m2 (including cut-off value), BMI= weight (kg)/height 2 (m2).

The investigator judged the subjects to be in good overall health based on their medical history, physical examination, vital signs, 12-lead electrocardiogram, laboratory tests (routine blood work, urine work, blood biochemistry, coagulation function), viral serology, and chest X-ray results (normal or abnormal test results have no clinical significance).

Fertile female subjects or male subjects who voluntarily signed ICF should be no fertile, sperm/egg donation for 6 months (female) or 90 days (male) from the beginning to the last dose, and voluntary use highly effective contraception (including partner) (non-drug contraception is required during the trial).

Fully understand the trial content and possible adverse reactions, have the ability to communicate with researchers normally, while complying with study requirements, follow protocol procedures and restrictions, and be able to visit on time.

Exclusion Criteria:

Subjects with a prior or present history of clinically abnormal metabolic, liver, kidney, hematological, pulmonary, cardiovascular, gastrointestinal, urinary, endocrine, neurological, or psychiatric disease who were judged by the investigator to be unsuitable for participation in this study.

Subjects with digestive tract disease or any condition that may affect drug absorption, such as a history of liver and gallbladder disease, gastrointestinal disease, gastrointestinal surgery (except appendectomy) or a history of chronic pancreatitis, idiopathic acute pancreatitis, or habitual diarrhea.

Allergic constitutions (such as allergies to two or more drugs, foods, and pollen), or determined by the investigator, may be allergic to the investigational product or any component of the investigational product.

Acute respiratory infections within 2 weeks before screening; Or have a history of fungal infection.

For patients with abnormal vital signs (blood pressure, pulse rate, ear temperature) and clinically significant results, the abnormal values of each vital sign are:Body temperature (ear temperature) >37.5 ℃; Systolic blood pressure (recumbent) <90 mmHg or ≥140 mmHg; Diastolic blood pressure (lying) <50 mmHg or ≥90 mmHg; Pulse rate (lying position) <50 beats/min or >100 beats/min.

QTcF interval > 450ms or < 300 ms (Fridericia's correction), or QRS>120ms. Abnormal liver function: alanyl aminotransferase (ALT) or aspartate aminotransferase (AST) higher than the upper limit of normal or serum total bilirubin (TBIL) greater than 1.5 times the upper limit of normal, who judged clinical significance by investigators.

Subjects estimate glomerular filtration rate <90 mL/min/1.73 m2. Subjects virus serological test (hepatitis B virus surface antigen, hepatitis C virus antibody, human immunodeficiency virus antibody, treponema pallidum specific antibody TPPA) positive results.

Subjects with a history of drug abuse (morphine, dimethylene dioxyamphetamine, methamphetamine, THC, ketamine, cocaine) or who screened positive for drug abuse.

Women who are pregnant or breastfeeding, or who test positive for blood pregnancy.

Subjects who have used any P-gp or CYP inducer or inhibitor within 30 days before screening, or any prescription or Chinese herbal medicine within 4 weeks before the start of the trial, or over-the-counter or health care products (including polyvalent cations and metal supplements, etc.) within 2 weeks before the start of the trial; It should have a longer time interval if the elimination half-life is longer-at least 5 elimination half-lives for the drug.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 18 (Actual)
Dates: Start 2023-08-28 (Actual); Primary Completion 2023-12-05 (Actual); Study Completion 2024-04-26 (Actual)

PRIMARY OUTCOMES:
PK parameters of active metabolite ZX-7101 in healthy Chinese adult subjects after a single oral ZX-7101A tablet combined with multiple oral oseltamivir phosphate capsules | Day1,Day2,Day3,Day5,Day10,Day15,Day20;Conbined period Day1,Day2,Day3,Day6,Day10,Day15,Day20
  Cmax
PK parameters of active metabolite ZX-7101 in healthy Chinese adult subjects after a single oral ZX-7101A tablet combined with multiple oral oseltamivir phosphate capsules | Day1,Day2,Day3,Day5,Day10,Day15,Day20;Conbined period Day1,Day2,Day3,Day6,Day10,Day15,Day20
  AUC0-t
PK parameters of active metabolite ZX-7101 in healthy Chinese adult subjects after a single oral ZX-7101A tablet combined with multiple oral oseltamivir phosphate capsules | Day1,Day2,Day3,Day5,Day10,Day15,Day20;Conbined period Day1,Day2,Day3,Day6,Day10,Day15,Day20
  AUC0-inf

CONTACTS AND LOCATIONS:
Locations (1):
- Peking University Third Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No